CLINICAL TRIAL: NCT06585696
Title: A Phase 3 Clinical Study to Evaluate the Efficacy and Safety of Botulinum Toxin Type A for Injection (CU-20101) Compared With A Single Treatment of Botox ® and Repeated Treatment of CU-20101 in Moderate to Severe Glabellar Striae
Brief Title: A Phase 3 Clinical Study to Evaluate the Efficacy and Safety of Botulinum Toxin Type A for Injection (CU-20101)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cutia Therapeutics（Wuxi）Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CU-20101-305
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Glabellar Frown Lines
Keywords: CU-20101

STUDY DESIGN:
Intervention Model Description: Parallel +Single Group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botox® (Active Comparator): CU-20101 treatment for Moderate to Severe Glabellar Striae
  Interventions: Drug: CU-20101 treatment for Moderate to Severe Glabellar Striae
- CU-20101 (Experimental): CU-20101 treatment for Moderate to Severe Glabellar Striae
  Interventions: Drug: CU-20101 treatment for Moderate to Severe Glabellar Striae

INTERVENTIONS:
Drug: CU-20101 treatment for Moderate to Severe Glabellar Striae — Part I (randomized double-blind controlled study) Study Part 1 consisted of a 1-day baseline/treatment period (randomized and received 1 dose of study treatment) and a 12-week post-treatment follow-up period.
  Part II (open-label study) For subjects who completed Part I of the study, they automatically entered Period 2 of the study. To evaluate the safety, efficacy, and immunogenicity of repeated injections of CU-20101 in the treatment of moderate to severe glabellar striae if they meet the criteria for repeat treatment (as shown in Figure 1, at least 12 weeks apart from each test drug injection). If repeat treatment criteria are not met at follow-up, follow-up may continue after 4 weeks until the next treatment is met. The last study treatment was no later than Day 253 ± 7 days (Week 36).

SUMMARY:
This is a Phase 3 clinical study to evaluate the efficacy, safety, and immunogenicity of single/repeated injections of CU-20101 in the treatment of moderate to severe glabellar lines. The study consisted of a 7-day screening period, Study Part 1 (randomized double-blind controlled study) and Period 2 (open-label study). Part I was a multicenter, randomized, double-blind, single-injection, active-drug parallel-controlled, non-inferiority design clinical study to evaluate the efficacy, safety, and immunogenicity of CU-20101 in the treatment of moderate to severe glabellar stria compared with a single injection of Botox®; part 2 was an open-label study to evaluate the efficacy, safety, and immunogenicity of repeated injections of CU-20101 in the treatment of moderate to severe glabellar lines.

DETAILED DESCRIPTION:
Part I (randomized double-blind controlled study) Study Part 1 consisted of a 1-day baseline/treatment period (randomized and received 1 dose of study treatment) and a 12-week post-treatment follow-up period. It is proposed to enroll 554 subjects with moderate to severe glabellar lines. Subjects eligible for inclusion were randomized in a 1: 1 ratio to CU-20101 or Botox® according to the stratification factors. Stratification factors were severity of glabellar lines at baseline (moderate vs. severe) when trying to frown as assessed on site by the investigator.

After completing the dosing of Part I and assessments of relevant examinations, subjects will return to the study site on Day 29 ± 7 days (Week 4), Day 57 ± 7 days (Week 8), and Day 85 ± 7 days (Week 12) for follow-up of efficacy, safety, and immunogenicity assessments (Figure 1).

Part II (open-label study) For subjects who completed Part I of the study, they automatically entered Period 2 of the study. To evaluate the safety, efficacy, and immunogenicity of repeated injections of CU-20101 in the treatment of moderate to severe glabellar striae if they meet the criteria for repeat treatment (at least 12 weeks apart from each test drug injection). If repeat treatment criteria are not met at follow-up, follow-up may continue after 4 weeks until the next treatment is met. The last study treatment was no later than Day 253 ± 7 days (Week 36).

Criteria for repeat therapy are (all of the following criteria must be met): 1.The severity of glabellar lines was assessed by the investigator on-site when the subject tried to frown, with an FWS score of 2 or 3 points; 2.The subjects self-assessed the severity of glabellar lines on the spot when they frowned with an FWS score of 2 or 3; 3.Meets the wishes of the subject; 4.All other inclusion criteria were met and none of the exclusion criteria were met.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria at the same time to be enrolled in the study:

  1. After being fully informed, fully aware of the content, process, benefits and possible adverse reactions of the study, and voluntarily participate in the study, and sign the informed consent form;
  2. Men or women aged 18-65 years (including boundary values);
  3. At screening, the investigator assessed the severity of glabellar lines when the subject tried to frown based on a 4-point FWS, with a score of ≥ 2 points;
  4. Subjects self-assessed the severity of glabellar lines when trying to frown based on a 4-point FWS score ≥ 2 points;
  5. Subjects were able to communicate well with the investigator and were willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Subjects who met any of the following exclusion criteria were not eligible for enrollment into the study:

  1. Subjects with skin abnormalities, including active infections (e.g., herpes simplex, acne, etc.), skin diseases (e.g., psoriasis, eczema, etc.), scars, etc., which may interfere with the study assessment as judged by the investigator;
  2. Subjects with diseases that may affect neuromuscular function (e.g., myasthenia gravis, Lambert-Easton syndrome, amyotrophic lateral sclerosis, etc.); or previous history of epilepsy;
  3. Previous history of facial paralysis and ptosis;
  4. Significant facial asymmetry;
  5. Physical stretching methods (e.g., manual stroking of equality) do not reduce eyebrow lines;
  6. Subjects allergic to the investigational product and its excipients (e.g., botulinum toxin, serum albumin, etc.);
  7. Subjects with prior surgery on the upper face (e.g. eyebrow lifting surgery), autologous fat implantation, semi-permanent or permanent material injection filling or implantation;
  8. Subjects who have received botulinum toxin injection of any serum type within 6 months prior to screening;
  9. Subjects who have received degradable fillers such as hyaluronic acid, collagen, etc. in the upper facial region within 12 months prior to screening;
  10. Subjects who have received intense pulsed light (photon), chemical denudation, etc., within 3 months prior to screening; for partial radiofrequency or high-energy laser treatment, the investigator should extend the interval to 6 months or more according to the actual situation;
  11. Subjects who plan to receive other medical aesthetic treatments (e.g., laser, injection tamponade, chemical peeling, etc.) or any treatment that may result in significant weight change (e.g. liposuction surgery, oral weight loss drugs, etc.) or who are expected to require treatment with botulinum toxin of any serum type (other than study intervention) during the study;
  12. Subjects taking oral retinoids within 6 months prior to screening or topical retinoids on the face within 3 months prior to screening;
  13. Subjects who have used the following systemic drugs within 1 month prior to screening: drugs with muscle relaxant effects (e.g., tubocurarine chloride, dantrolene sodium, baclofen, etc.), aminoglycoside antibiotics (e.g., gentamicin sulfate, neomycin sulfate, etc.), polypeptide antibiotics (e.g., polymyxin B sulfate), tetracycline antibiotics, lincolamides, anticholinergic drugs (e.g., hyoscine butylbromide hydrochloride, benzhexol hydrochloride, etc.), benzodiazepines (e.g., etizolam, etc.), benzamide drugs (e.g., thiopride hydrochloride, sulpiride, etc.);
  14. Subjects who have used anticoagulants or non-steroidal anti-inflammatory drugs within 7 days prior to study drug administration; for menstruating subjects, the study drug injection may be delayed as needed to avoid the menstrual period;
  15. Pregnant or lactating women;
  16. Male or female subjects unwilling to use reliable contraception throughout the trial (except female subjects of non-childbearing potential);
  17. According to vital signs, physical examination, 12-lead electrocardiogram, laboratory tests (hematology, blood biochemistry, urinalysis, coagulation) and blood pregnancy test at screening, the investigator judged the abnormalities as clinically significant and assessed as not suitable for participation in the investigator;
  18. Positive results of any test result for hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody and treponema pallidum antibody;
  19. Participation in any clinical trial as a subject within 30 days prior to screening;
  20. Subjects with psychiatric disorders that may affect the conduct of the study as judged by the investigator;
  21. Previous history of drug or drug abuse;
  22. Subjects who are in the acute phase of disease at screening, or have serious systemic diseases, etc., and are judged by the investigator to be ineligible for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-11-20 (Actual)

PRIMARY OUTCOMES:
• Proportion of subjects with an FWS score of 0 or 1 and both with a decrease of ≥ 2 points from baseline as assessed on-site by the investigator and the subject at Week 4 after the first round of injection. | Stage 1: Screening period of 7 days, treatment + follow-up about 12 weeks, the longest 92 days; Stage 2: Treatment + follow-up for about 36 weeks. All together takes up to 344 days
  • Proportion of subjects with an FWS score of 0 or 1 and both with a decrease of ≥ 2 points from baseline as assessed on-site by the investigator and the subject at Week 4 after the first round of injection.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wu, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No